CLINICAL TRIAL: NCT03604315
Title: Serial Imaging of the Novel Radiotracer [^18F] FLuorthanatrace ([^18F] FTT) by PET/CT
Brief Title: Serial Imaging of the Novel Radiotracer [^18F] FLuorthanatrace ([^18F] FTT) by PET/CTF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0319; NCI-2018-01137 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0319 (Other: M D Anderson Cancer Center); R01CA249329 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma; Fallopian Tube Carcinoma; Ovarian Carcinoma; Primary Peritoneal Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (FDG PET/CT, [18F]FTT PET/CT) (Experimental): Patients receive FDG IV and undergo FDG PET/CT scan over 20-30 minutes if they have not already had one per standard of care. At least 20-24 hours later, patients receive fluorine F 18 fluorthanatrace IV and undergo [18F]FTT PET/CT over 1 hour.
  Interventions: Procedure: Computed Tomography; Radiation: Fludeoxyglucose F-18; Radiation: Fluorine F 18 Fluorthanatrace; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo FDG PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Computed Tomography — Undergo [18F]FTT PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Radiation: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: Fluorine F 18 Fluorthanatrace — Given IV
  Other Names: [18F]FluorThanatrace; [18F]FTT
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Procedure: Positron Emission Tomography — Undergo [18F]FTT PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies how well fluorine F 18 fluorthanatrace positron emission tomography (PET)/computed tomography (CT) works in patients with solid tumors. Fluorine F 18 fluorthanatrace is a radioactive tracer, a type of imaging agent that is labeled with a radioactive tag and injected into the body to help with imaging scans. PET/CT uses a scanner to make detailed, computerized pictures of areas inside the body. PET/CT with Fluorine F 18 fluorthanatrace may allow more tumor cells to be found in patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

- Evaluate fluorine F 18 fluorthanatrace ([18F]Fluorthanatrace) positron emission tomography/computed tomography (PET/CT) as an imaging biomarker of poly [ADP-ribose] polymerase (PARP)-1 activity in 3 cohorts of cancer patients: 1) ovarian, fallopian tube, primary peritoneal 2) breast cancer, and 3) non-ovarian, non-breast solid tumor.

SECONDARY OBJECTIVES:

* Evaluate the safety of [18F]Fluorthanatrace.
* Correlate [18F]Fluorthanatrace uptake measures with BRCA mutation status.
* Correlate [18F]Fluorthanatrace uptake measures with poly [ADP-ribose] polymerase (PARP-1) activity in tumor tissue samples in patients who undergo biopsies.
* Evaluate change in [18F]Fluorthanatrace uptake measures after therapy initiation with repeat imaging before and after treatment initiation.
* To confirm the variability of imaging findings from repeated [18F]FTT PET/CT over 1 week before treatment initiation
* Determine the change in [18F]FluorThanatrace uptake before treatment initiation and at time of clinical progression
* Correlate [18F]FluorThanatrace uptake at time of clinical progression measures with genetic reversion mutation status

OUTLINE:

Patients receive fluorodeoxyglucose (FDG) intravenously (IV) and undergo FDG PET/CT scan over 20-30 minutes if they have not already had one per standard of care. At least 20-24 hours later, patients receive fluorine F 18 fluorthanatrace IV and undergo fluorine F 18 fluorthanatrace ([18F]FTT) PET/CT over 1 hour.

After completion of study treatment, patients are followed up at 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* History of known or suspected solid tumor.
* At least one lesion ≥ 1.0 cm that is seen on standard imaging (e.g. computed tomography [CT], magnetic resonance imaging [MRI], ultrasound, fludeoxyglucose [FDG] PET/CT).

Exclusion Criteria:

* Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential < 2 weeks prior to screening as standard of care.
* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.
* Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Poly (ADP-ribose) polymerase inhibitor (PARP)-1 activity as assessed by fluorine F 18 fluorthanatrace positron emission tomography/computed tomography | Up to 4 years
  Data will be generated for semi-parametric uptake of both tracers by patient and by lesion as well as by PARP activity, and summarized as mean and standard deviation (SD) across patients. For patients for whom tumor tissue is saved, the correlation of uptake values and PARP activity as assayed from biopsy specimens will be measured using the rank correlation (Spearman's rho), and test for significance compared to no correlation.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 4 years
BRCA mutation status | Up to 4 years
  To determine any correlation with BRCA status, fluorine F 18 fluorthanatrace ([18F]FTT) uptake values (mean and SD) across patient and lesion (summing across lesions) will be summarized, by BRCA status group. Group difference will be tested using t-tests.
PARP-1 activity in tumor tissue samples | Up to 4 years
  Data will be generated for semi-parametric uptake of both tracers by patient and by lesion as well as by PARP activity, and summarized as mean and SD across patients. For patients for whom tumor tissue is saved, the correlation of uptake values and PARP activity as assayed from biopsy specimens will be measured using the rank correlation (Spearman's rho), and test for significance compared to no correlation.
Change in fluorine F 18 fluorthanatrace uptake measures after therapy | Baseline up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Lilie L Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lin LL, Wong F, Lin R, Yap T, Litton JK. Pharmacodynamic Activity of [18F]-Fluorthanatrace Poly(ADP-ribose) Polymerase Positron Emission Tomography in Patients With BRCA1/2-Mutated Breast Cancer Receiving Talazoparib. JCO Precis Oncol. 2024 Aug;8:e2400303. doi: 10.1200/PO.24.00303. PMID 39208372
- See also: MD Anderson Cancer Center — http://www.mdanderson.org